CLINICAL TRIAL: NCT04611334
Title: Effects of Heart Rate Variability Biofeedback to Improve Automatic Nervous Function, Inflammatory Response, Physiological and Psychological Symptom Distress in Patients With Chronic Kidney Disease：A Randomized Control Trial
Brief Title: The Effects of HRV Biofeedback on Chronic Kidney Disease Patient.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yu-Ju Chen, Dean of nursing, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1-2020-9-20
Record Dates: First submitted 2020-09-26; First posted 2020-11-02 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Autonomic Dysfunction; Inflammatory Response; Chronic Kidney Diseases
MeSH Terms: conditions — Primary Dysautonomias; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): HRV biofeedback
  Interventions: Behavioral: heart rate variability biofeedback
- control group (No Intervention): routine care

INTERVENTIONS:
Behavioral: heart rate variability biofeedback — Heart rate variability biological feedback training is carried out in the outpatient meeting room of the hospital, including once a week, 30 minutes of hospital training each time, using Medea physiological feedback device portable Bluetooth physiological signal Feedback system (Medical Device Input No. 027390). Designed as two stages, stage one (the first week) first teaches the subject how to perform abdominal breathing, and connects the physiological feedback device to monitor the patient's breathing and heart rate changes, and sets the breath per minute according to the subject's resonance frequency . Stage two (second-four weeks) guide the case to understand the resonance relationship between breathing and heart rate, and then achieve the effect of matching heart and breath. It is also equipped with a pressure relief device (Helico Inc., New York, NY, USA) for self-practice at home.
  Arms: experimental group

SUMMARY:
The prevalence and incidence of end-stage renal disease in Taiwan ranks highest in the world, and it is based on the 2018 health welfare According to statistics from the Ministry of Foreign Affairs, kidney disease is the ninth leading cause of death in Taiwan. As the course of chronic kidney disease (CKD) progresses, autonomic nervous system dysfunction, inflammation, and physical and psychological symptoms (such as fatigue, sleep disturbance, and depression) will increase, which will further damage the structure and function of the kidney Intensified, increasing the demand for dialysis treatment and the risk of cardiovascular disease, which consumes social and medical costs. If the investigators can intervene in a feasible measure to effectively regulate the autonomic nervous function of CKD patients, reduce inflammation and physical and psychological symptoms, and delay the progression of the disease, it will be the main goal of caring for CKD patients. To explore the intervention of heart rate variability biofeedback, which can improve the autonomic nervous function (heart rate variability [Heart Rate Variability]), inflammatory response (interleukin-6 [Interleukin-6, IL-6], C-reactive protein [ C reaction protein, CRP]) and physical and psychological symptoms (such as reducing fatigue, sleep disturbance and depression).

DETAILED DESCRIPTION:
This study adopts an experimental research design and convenient sampling method. It is accepted in the nephrology clinic of a northern medical center in Taiwan. It is estimated that 80 patients will be enrolled. After the patients have signed the consent form, use the sealed envelope website (http://www.sealedenvelope.com) will randomly assigned to the experimental group and the control group. The experimental group receive HRV biofeedback for four consecutive weeks, combined with eight-week StressEraser home practice; the control group received general routine care. Both groups of cases were repeated three times on the day of acceptance, one month and three months after the case were accepted, a total of three repeated measurements of physiological indicators (HRV, IL-6, CRP) and symptom scales (Piper Fatigue Scale, Chinese version of Pittsburgh Sleep Quality Table, the second edition of the Chinese version of the Baker Depression Scale) to evaluate the effectiveness of HRV biofeedback. The research results will be statistically analyzed with SPSS version 23.0, and with descriptive statistics, the distribution of basic demographic data and the measurement results of various indicators will be analyzed. Paired-sample t-test, independent-sample t-test, and multivariate analysis of variance (MANOVA) were used to analyze the statistical results of intervention effectiveness inference; the significance level was set to 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of chronic kidney disease
2. Clear consciousness
3. able to communicate in Mandarin or Taiwanese
4. no urgency in the past three months
5. No hospitalization record in the past three months.

Exclusion Criteria:

1. arrhythmia
2. with pacemaker
3. those with visual or hearing impairments that cannot be corrected and hinder communication
4. receiving dialysis treatment
5. receiving kidneys Transplant recipients
6. history of rheumatic immune disease or cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-11-18 (Estimated); Study Completion 2023-12-18 (Estimated)

PRIMARY OUTCOMES:
autonomic nerve function | baseline
  heart rate variability index
autonomic nerve function | 1 month
  heart rate variability index
autonomic nerve function | 3 month
  heart rate variability index

SECONDARY OUTCOMES:
inflammatory response 1 | baseline
  C reaction protein, CRP(ng/ml)
inflammatory response 2 | baseline
  Interleukin-6, IL-6(pg/ml)
inflammatory response 1 | 1 month
  C reaction protein, CRP(ng/ml)
inflammatory response 2 | 1 month
  Interleukin-6, IL-6(pg/ml)
inflammatory response 1 | 3 month
  C reaction protein, CRP(ng/ml)
inflammatory response 2 | 3 month
  Interleukin-6, IL-6(pg/ml)
symptom distress(fatigue) | baseline
  Piper fatigue scale(Chinese version): Likert's four-point quantitative scale is scored, calculated on a scale of 0-3, with a total score of 0-48. The higher the score, the more serious the fatigue.
symptom distress(sleep) | baseline
  Pittsburgh Sleep Quality Index
symptom distress(depression) | baseline
  Beck Depression Inventory-II
symptom distress(fatigue) | 1 month
  Piper fatigue scale(Chinese version): Likert's four-point quantitative scale is scored, calculated on a scale of 0-3, with a total score of 0-48. The higher the score, the more serious the fatigue.
symptom distress(sleep) | 1 month
  Pittsburgh Sleep Quality Index
symptom distress(depression) | 1 month
  Beck Depression Inventory-II
symptom distress(fatigue) | 3 month
  Piper fatigue scale(Chinese version): Likert's four-point quantitative scale is scored, calculated on a scale of 0-3, with a total score of 0-48. The higher the score, the more serious the fatigue.
symptom distress(sleep) | 3 month
  Pittsburgh Sleep Quality Index
symptom distress(depression) | 3 month
  Beck Depression Inventory-II

CONTACTS AND LOCATIONS:
Overall Officials: YU-CHAN LIN, master, Principal Investigator — Tri-Service Medical Center Nurse; CHIA-PEI Chen, Principal Investigator — Graduate Student
Locations (1):
- Tri-Service Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No